CLINICAL TRIAL: NCT02838004
Title: An Open Label, Non-comparative Study to Assess the Visual Performances and Safety of a Progressive Multifocal Intraocular Lens With Extended Depth of Focus
Brief Title: Non-comparative Study to Assess the Visual Performances and Safety of a Progressive Multifocal Intraocular Lens
Acronym: PSM15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SIFI SpA (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PSM15
Record Dates: First submitted 2016-07-12; First posted 2016-07-20 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Cataract; Presbyopia
Keywords: Refractive lens exchange (RLE) or cataract surgery
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm receiving Mini WELL Ready IOL (Experimental): IOL implantation for cataract
  Interventions: Device: IOL MINI WELL READY

INTERVENTIONS:
Device: IOL MINI WELL READY — IOL MINI WELL READY

SUMMARY:
This is an interventional, non-controlled, multicenter international trial with a prospective design on one cohort of patients.

DETAILED DESCRIPTION:
To evaluate if the positive results (to assure a good visual acuity at all distances and a good quality of life in terms of glasses independence and absence of undesired events), obtained experimentally using the IOL MINI WELL READY, can be confirmed in the practical surgical routine with a population belonging to different EU countries

ELIGIBILITY:
Inclusion Criteria:

* Any gender and age above 18 years.
* Refractive lens exchange (RLE) or cataract surgery.
* Healthy corneas, not treated surgically.
* Patients willing to have surgery in both eyes in a short period of time (within 2 weeks).
* Patients request to receive the IOL MINI WELL READY implant

Exclusion Criteria:

* Previous corneal surgery (i.e. pterygium, refractive surgery).
* Eye diseases determining a probable postoperative visual acuity < 20/40.
* Pseudoexfoliation.
* Abnormal pupil size and position.
* Use of contact lens 30 days before the preoperative visit.
* Corneal warpage.
* Predicted postoperative corneal astigmatism higher than 1 D.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
UDVA (Uncorrected Distance Visual Acuity) | 30 days
  Visual acuity mesurement

SECONDARY OUTCOMES:
Adverse Device Effects (ADE); Serious Adverse Device Effects (SADE); Unexpected Serious Adverse Device Effects (USADE); Adverse Events (AE); Serious Adverse Events (SAE). | 4 months
  Safety assessment

OTHER OUTCOMES:
Visual Acuity Evaluation | 4 months
  Corrected Distance Visual Acuity (CDVA)
Visual Acuity Evaluation | 4 months
  Uncorrected Near Visual Acuity (UNVA)
Visual Acuity Evaluation | 4 months
  Distance-Corrected Near Visual Acuity (DCNVA)
Visual Acuity Evaluation | 4 months
  Corrected Near Visual Acuity (CNVA)
Visual Acuity Evaluation | 4 months
  Uncorrected Intermediate Visual Acuity (UIVA)
Visual Acuity Evaluation | 4 months
  Distance-Corrected Intermediate Visual Acuity (DCIVA)
Halos and Glare evaluation | 4 months
  Onset of halos Onset of glare during night vision
Contrast sensitivity | 4 months
  Contrast sensitivity, at 3 meters, under photopic conditions and with the correction for distance, using YANG SMART (SIFI Medtech), with sine wave gradings (''vistech")
Reading Performance | 4 months
  Reading Performance tested with Radner Reading Chart - Precision Vision:
  The test will be performed from the largest to the smallest size of letters in two sessions:
  * Binocular, without the correction for distance, at 40 cm
  * Binocular, with the correction for distance, at 40 cm
Defocus Curve | 4 months
  Binocular defocus curves with step of 0.5 D (from +2.0 to -5.0 D) under photopic conditions.

CONTACTS AND LOCATIONS:
Overall Officials: GERD U. AUFFARTH, Prof. Dr., Principal Investigator — RUPRECHT KARLS UNIVERSITATS AUGENKLINIK HEIDELBERG
Locations (1):
- Prof.Dr. Gerd U. Auffarth, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang T, Jiang J, Zhou Y, Zhao GQ, Li H, Zhao SY. Cataract surgery in aged patients: phacoemulsification or small-incision extracapsular cataract surgery. Int J Ophthalmol. 2011;4(5):513-8. doi: 10.3980/j.issn.2222-3959.2011.05.11. Epub 2011 Oct 18. PMID 22553713
- [Background] Packer M, Fine IH, Hoffman RS. Aspheric intraocular lens selection: the evolution of refractive cataract surgery. Curr Opin Ophthalmol. 2008 Jan;19(1):1-4. doi: 10.1097/ICU.0b013e3282f2d791. No abstract available. PMID 18090888
- [Background] Kohnen T, Klaproth OK, Buhren J. Effect of intraocular lens asphericity on quality of vision after cataract removal: an intraindividual comparison. Ophthalmology. 2009 Sep;116(9):1697-706. doi: 10.1016/j.ophtha.2009.03.052. Epub 2009 Jul 29. PMID 19643497
- [Background] Lehmann R, Waycaster C, Hileman K. A comparison of patient-reported outcomes from an apodized diffractive intraocular lens and a conventional monofocal intraocular lens. Curr Med Res Opin. 2006 Dec;22(12):2591-602. doi: 10.1185/030079906X158039. PMID 17166341
- [Background] Leyland M, Zinicola E. Multifocal versus monofocal intraocular lenses in cataract surgery: a systematic review. Ophthalmology. 2003 Sep;110(9):1789-98. doi: 10.1016/S0161-6420(03)00722-X. PMID 13129879
- [Background] Steinert RF. Visual outcomes with multifocal intraocular lenses. Curr Opin Ophthalmol. 2000 Feb;11(1):12-21. doi: 10.1097/00055735-200002000-00004. PMID 10724823
- [Background] Munoz G, Albarran-Diego C, Ferrer-Blasco T, Sakla HF, Garcia-Lazaro S. Visual function after bilateral implantation of a new zonal refractive aspheric multifocal intraocular lens. J Cataract Refract Surg. 2011 Nov;37(11):2043-52. doi: 10.1016/j.jcrs.2011.05.045. PMID 22018366
- [Background] Ucakhan OO, Ozkan M, Kanpolat A. Anterior chamber parameters measured by the Pentacam CES after uneventful phacoemulsification in normotensive eyes. Acta Ophthalmol. 2009 Aug;87(5):544-8. doi: 10.1111/j.1755-3768.2008.01305.x. Epub 2008 Sep 11. PMID 18786130
- [Background] Savini G, Olsen T, Carbonara C, Pazzaglia S, Barboni P, Carbonelli M, Hoffer KJ. Anterior chamber depth measurement in pseudophakic eyes: a comparison of Pentacam and ultrasound. J Refract Surg. 2010 May;26(5):341-7. doi: 10.3928/1081597X-20090617-02. Epub 2010 May 19. PMID 20506991
- [Background] Attia MS, Khoramnia R, Auffarth GU, Kirchner M, Holzer MP. Near and intermediate visual and reading performance of patients with a multifocal apodized diffractive intraocular lens using an electronic reading desk. J Cataract Refract Surg. 2016 Apr;42(4):582-90. doi: 10.1016/j.jcrs.2015.11.047. PMID 27113882
- [Background] Maxwell WA, Cionni RJ, Lehmann RP, Modi SS. Functional outcomes after bilateral implantation of apodized diffractive aspheric acrylic intraocular lenses with a +3.0 or +4.0 diopter addition power Randomized multicenter clinical study. J Cataract Refract Surg. 2009 Dec;35(12):2054-61. doi: 10.1016/j.jcrs.2009.06.041. PMID 19969208